CLINICAL TRIAL: NCT05627583
Title: Τhe Effect of Nutritional rEhabilitation in Patients With Anorexia Nervosa on Markers Associated With Disease severiTy
Brief Title: Nutritional Rehabilitation and Markers of Severity in Anorexia Nervosa
Acronym: EAT
Status: Completed | Type: Observational
Sponsor: Harokopio University (Other)
Collaborators: National and Kapodistrian University of Athens (Other); Sismanoglio General Hospital (Other); Attikon Hospital (Other); National Hellenic Research Foundation (Other)
Responsible Party: Principal Investigator, Andriana C. Kaliora, Prof. in Human Nutrition and Foods, Harokopio University
Other Study IDs: EAT study
Record Dates: First submitted 2022-11-08; First posted 2022-11-25 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2024-10

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa | interventions — Rehabilitation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Fecal samples are used to extract DNA for NGS
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Anorexia Nervosa (AN): Anorexia Nervosa patients hospitalized for rehabilitation
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Rehabilitation — Hospitalized patients with AN under treatment for rehabilitation

SUMMARY:
The design of this project is a longitudinal trial in patients with Anorexia Nervosa (AN) during in-hospital rehabilitation. Τhe structure of the study, the questionnaires and data protection policy prepared exclusively for our study, have been reviewed and standardised at Institutional Review Boards (Ethics Committees, IRBs,) in Harokopio University of Athens (HUA), Eginition Hospital (EH), Attiko Hospital (AH) and Sismanoglio Hospital (SG).

AN is a psychiatric disorder followed by a psychopathologic concerning of body image and very low body weight due to extreme self-starvation. The exact pathogenesis of AN remains unknown with neurobiological, gastrointestinal, neuroendocrinological, immunological, and genetic factors suspected to be implicated. Furthermore, many metabolic traits, biochemical, biological or/and anthropometrical, are manifested during the maintaining effort of patients to achieve lower body weight. Self-inflicted starvation is the primary and essential causation of the pathological outcomes of the disorder. These outcomes involve all biological systems and organs. The role of the immune system in AN is critical as levels of pro-inflammatory cytokines are increased and the immune system is dysregulated. Other contributors to AN pathogenesis have been proposed, such as increased oxidative stress, dysbiosis of the gut microbiota and altered metabolomic profiles. Treatment options for patients with AN constitutes outpatient and inpatient care accordingly with the severity of the disorder. So far, no biomarker has been strongly proposed as an indicator of the disorder's severity or for assessing the progression of the treatment.

The purpose of this study is to assess and monitor the nutritional rehabilitation of patients with AN during hospitalization treatment. Throughout the treatment's course, nutrition and feeding process, vital signs, psychopathology and biological samples will be gathered and statistical analysis of these data is expected to reveal potential biomarker/s for monitoring the progression of recovery.

DETAILED DESCRIPTION:
Inpatients with AN and non-eating disorders control subjects will be informed about the project outline, objectives and inclusion criteria.

Monitoring of AN patients will take place during in-hospital rehabilitation. Physical exam, lab tests, bioelectrical impedance analysis and psychometric evaluation will take place twice a month. Plasma and serum will be collected and isolated form blood samples, while stool samples will be collected for Nuclear Magnetic Resonance (NMR) metabolomics analysis and in StoolFix tubes for DNA isolation from intestinal microbiota. For serum and plasma isolation, whole blood will be directly and properly drawn into a vacutainer tube and promptly centrifuged. Then, samples will be stored at -80C until further elaboration. Case record forms will be carefully checked for missing data and inconsistencies prior to developing a proper database based on data entry. The highest ethical standards and data protection will be considered.

Assessment will include Medical history, Anthropometric measurements, Vital signs, Nutrition, Subjective Global Assessment-Patient Generated (SGA-PG), Biochemical parameters, Appetite hormones, Inflammation markers, Oxidative stress markers, Composition of intestinal microbiota, Psychometric scales-measurements, Eating Attitude Test-26 (EAT-26), Eating Disorder Examination Questionnaire (EDE-Q), Spielberger State-Trait Anxiety Inventory (STAI), Beck Depression Inventory (BDI), Body Appreciation Scale (BAS), Sense of Coherence Scale (SOC), Visual Analogue Scale (VAS) for subjective appetite estimation

ELIGIBILITY:
Inclusion Criteria:

• Patients with Anorexia Nervosa according to the DSM-V (American Psychiatric Association, 2013)

Exclusion criteria:

• Antibiotic treatment before and during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 13 Males and females with AN who are hospitalized for rehabilitation
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-10-24 (Actual); Study Completion 2023-12-24 (Actual)

PRIMARY OUTCOMES:
Increase in Body Weight | Up to three months during inpatient rehabilitation
  Increase in body weight as a marker of rehabilitation

SECONDARY OUTCOMES:
Metabolic recovery in patients with AN | Up to three months during inpatient rehabilitation
  This study aims to investigate metabolic changes in the gut microbiome of patients with Anorexia Nervosa during nutritional rehabilitation. Stool samples will be collected at multiple time points throughout the in-hospital rehabilitation period. Metabolite concentrations will be analyzed using Nuclear Magnetic Resonance (NMR)-based metabolomics to assess longitudinal alterations associated with metabolic recovery.
Changes in ghrelin levels | Up to three months during inpatient rehabilitation
  As a marker of appetite ghrelin blood levels are measured.
Changes in blood metals and metalloids | Up to three months during inpatient rehabilitation
  Different metals and metalloids in plasma are evaluated applying ICP-MS.
Changes in leptin levels | Up to three months during inpatient rehabilitation
  Changes in leptin levels
Changes in IL-6 levels | Up to three months during inpatient rehabilitation
  Changes in IL-6 levels
Changes in serum oxidisability | Up to three months during inpatient rehabilitation
  Changes in serum oxidisability
Changes in EDE-Q | Up to three months during inpatient rehabilitation
  The EDE-Q is a marker of disorder severity.
Changes in EAT-total | Up to three months during inpatient rehabilitation
  EAT-total is a marker of disorder severity.

CONTACTS AND LOCATIONS:
Overall Officials: Andriana C. Kaliora, Study Director — Harokopio University
Locations (1):
- Kaliora, Andriana C., Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No